CLINICAL TRIAL: NCT00963222
Title: The Study of the Effects of Vitamin A Supplementation on Immune System and Th1/Th2 Balance in Patients With Atherosclerosis
Brief Title: The Study of the Effects of Vitamin A on Immune System in Patients With Atherosclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 86-04-27-6617
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Coronary Artery Disease; Vitamin A; CD4-Positive T-Lymphocytes; Th1 Cells; Th2 Cells
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- with atherosclerosis/ vitamin A (Active Comparator): patients with angiographically confirmed CAD (defined as luminal stenosis ≥50% in at least one major coronary artery branch)who receive 25000 IU/day vitamin A
  Interventions: Drug: vitamin A
- with atherosclerosis/ placebo (Placebo Comparator): patients with angiographically confirmed CAD (defined as luminal stenosis ≥50% in at least one major coronary artery branch)who receive placebo
  Interventions: Drug: placebo
- without atherosclerosis/ vitamin A (Active Comparator): patients in whom significant (e.g. stenosis ≥ 50%) CAD is ruled out by coronary angiography, who receive 2500 Iu/day vitamin A
  Interventions: Drug: vitamin A
- without athrosclerosis/ placebo (Placebo Comparator): patients in whom significant (e.g. stenosis ≥ 50%) CAD is ruled out by coronary angiography, who receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin A — 1 cap vitamin A 25000 IU/day for 3 month
  Arms: with atherosclerosis/ vitamin A; without atherosclerosis/ vitamin A
Drug: placebo — 1 cap placebo/day for 3 month
  Arms: with atherosclerosis/ placebo; without athrosclerosis/ placebo

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with 25000 IU preformed vitamin A (retinyl palmitate) or placebo for 3 months on immune system and Th1/Th2 balance in patients with and without atherosclerosis (documented with angiography).

DETAILED DESCRIPTION:
Atherosclerosis, the leading cause of death and disability in the world, is considered an inflammatory disease with a complex etiology. The immune system has a prominent role in the formation, development and destabilization of atherosclerotic plaques. A whole range of identified cytokines have been shown to play a part in atherogenesis, some with proatherogenic properties while others having antiatherogenic properties. With increasing evidence for the significant role of inflammation and the cytokines involved together with the Th1/Th2 imbalance in atherosclerosis and its progression to Coronary artery diseases (CADs), the control of cytokine production may become potential therapeutic targets and modulation of the Th1/Th2 balance may provide a new pharmacological tool to treat this disease. Vitamin A (VA) or VA-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. high level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid inhibits IL 12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or retinoic acid (RA) decreases IFNγ and increases IL5, IL10, and IL4 production. Thus, vitamin A deficiency biases the immune response in a Th1 direction, whereas high level dietary vitamin A may bias the response in a Th2 direction.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for enrollment of the patients and control subjects is consecutive patients of both sexes referred to the Division of Cardiology of the one of the Hospitals of Tehran University of Medical Sciences for coronary angiography for investigation of chest pain and/or suspected CAD.

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* Patients who have allergy to vitamin A compounds, OR
* Patients who have used vitamin supplements in last 3 months.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Serum levels of IL4, IL10, IFN γ, IL2, IL12 | first day and after 3 month
PBMC supernatant levels of IL4, IL10, IFN γ, IL2, IL12 | first day and after 3 month

SECONDARY OUTCOMES:
serum Total cholesterol | first day and after 3 month
serum HDL cholesterol | first day and after 3 month
serum triglycerides level | first day and after 3 month
serum Apo A, Apo B and CRP levels | first day and after 3 month
serum oxLDL | first day and after 3 month
RBP/ TTR ratio | first day and after 3 month
lymphocyte proliferation assay (MTT) | first day and after 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akbar saboor Yaraghi, PhD, Study Chair — Tehran University of Medical Sciences; Maryam Mahmoudi, MD, PhD student, Principal Investigator — Tehran University of Medical Siences; Fereidon Siassi, PhD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, School of Public Health, Tehran, Tehran Province, Iran